CLINICAL TRIAL: NCT03682861
Title: Effect of Glycogen Replenishment on Time Trial Performance Following a Glycogen Lowering Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor, Western University, Canada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 112747
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Carbohydrate Metabolism

STUDY DESIGN:
Intervention Model Description: It is a repeated measure design where each participant will undergo all four treatment in a randomized fashion to prevent any order effect. Treatments (recovery drinks) include a placebo which will be similar in taste and flavour to other treatments and three carbohydrate containing drinks mixed in water at different concentrations. Design of the study is composed of three main stages: 1) glycogen lowering exercise, 2) glycogen replenishment and rest and 3) performance based, timed cycling exercise. All participants will arrive fasted to the laboratory, performing an exercise protocol that lowers their glycogen levels, followed by ingestion of different drinks (every 30 min) during 2 hours of a 4 hour rest and finally performing a 20 km stationary bike test for the time to finish to evaluate the effect of recovery drinks ingested.
Who Masked: Participant
Masking Description: Flavoured water placebo drink with no energy or carbohydrate drinks in opaque bottles to keep participant blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo flavored drink similar to treatments but with no energy will be ingested post glycogen lowering exercise, followed by a 20 km time trial intervention
  Interventions: Behavioral: 20 km time trial performance; Behavioral: Glycogen lowering exercise
- Carbohydrate drinks (Experimental): Sweet corn derived starch mixed in water at three different concentrations (6%, 12% and 18%) will be ingested post glycogen lowering exercise, followed by a 20 km time trial intervention
  Interventions: Behavioral: 20 km time trial performance; Behavioral: Glycogen lowering exercise

INTERVENTIONS:
Behavioral: 20 km time trial performance — 20 km time trial cycling test will be conducted to measure the effect of different drinks on time
Behavioral: Glycogen lowering exercise — Glycogen will be lowered using a 10-min warm-up period at a workload of 50% max wattage power output (Wmax). Thereafter, participants will be instructed to cycle 2-min block periods at alternating workloads of 90% and 50% of Wmax, respectively. This will be continued until the participants are no longer able to complete the 2 min at 90% Wmax. That moment will be defined as the time at which the individual is unable to maintain cycling speed at 60 revolutions/min. At that moment the high-intensity block will be reduced to 80% Wmax. Again, athletes will cycle until they are unable to complete a 2-min block at 80% Wmax, after which the high-intensity block will be reduced to 70% Wmax. Finally, participants will be allowed to stop when pedalling speed could not be maintained at 70% Wmax.

SUMMARY:
Fifteen endurance-trained male/female will be randomly assigned to do four exercise and nutrition trials involving ingestion of four different concentrations of sweet corn derived starch (food component) in water (0, 1, 1.5 and 2 g. kg-1. h-1). Each trial will be separated by at least one week. During these four experimental trials athletes will be subjected to a glycogen-lowering cycling exercise protocol followed by a 4-h post-exercise recovery period (2h feeding then 2 hours of rest). At the end of 4-h period they will do a 20 kilometre time trial test on a stationary bike in a laboratory condition to measure the effect of different glycogen repletion rates on exercise performance.

DETAILED DESCRIPTION:
Post-exercise glycogen synthesis rate is an important factor in determining the time needed to recover. Glycogen synthesis is affected not only by the extent of glycogen depletion but also in a more direct manner by the type, duration, and intensity of the preceding exercise because these will differentially influence the acute enzymatic changes as well as recovery from the acute changes that are induced by strenuous exercise. To optimize glycogen synthesis rates, adequate amounts of carbohydrate should be ingested. It has been suggested initially that a carbohydrate intake of 0.35 g·kg body wt-1 ·h-1 , provided at 2-h intervals, maximized muscle glycogen synthesis. Others observed no differences in glycogen storage rates after subjects ingested 0.75 or 1.5 g carbohydrate·kg-1 · h-1 provided at 2-h intervals. In a follow-up study, it was reported that an intake of >0.5 g·kg-1 · h-1 is necessary to maximize post-exercise glycogen synthesis if supplements are administered at 2-h intervals. Higher glycogen synthesis rates have been reported in studies in which carbohydrates were ingested more frequently and at higher ingestion rates than in previous studies. Other efforts to increase glycogen synthesis rates by changing the form of administration (ie, as a solution, as a solid, or intravenously) have been unsuccessful. While the above range of intake rates has been suggested to maximize muscle glycogen resynthesis post-exercise, the required dosage with sweet corn derived high glycemic starch and its effect on a subsequent time trial exercise is currently unknown. So, investigators objective in this experiment is to find out optimal sweet corn derived recovery ingestion dose by using a glycogen lowering exercise protocol, followed by glycogen repletion via ingestion and a subsequent 20 km time trial cycling performance.

ELIGIBILITY:
Inclusion Criteria:

* are a healthy male or female endurance athlete of 18- 40 years of age
* have ≥2 y endurance training experience; training for ˃1 h/day

Exclusion Criteria:

* Have symptoms or take medication for respiratory disease
* Have symptoms or take medication for cardiovascular disease
* Have symptoms or take medication for metabolic disease
* Have symptoms or take mediation for neuromuscular disease
* Use heart rate or blood pressure medications
* Use any medications with side effects of dizziness, lack of motor control, or slowed reaction time
* Have any cardiovascular or neuromuscular limitations to exercise
* Are pregnant or find out that you are pregnant during experiment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
20 km time trial | 40 minutes
  participants will ride for 20 km on a stationary bike and time to finish will be measured

SECONDARY OUTCOMES:
VO2 | 2 hours
  VO2 will be measured using a metabolic cart
Blood glucose | 2 hours
  glucose will be measured using glucometer
VCO2 | 2 hours
  VCO2 will be measured using a metabolic cart
Serum insulin | 2 hours
  Insulin will be measured using an immumoassay kit
Blood lactate | 2 hours
  blood lactate will be measured using lactate meter

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory (Western University), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ivy JL. Glycogen resynthesis after exercise: effect of carbohydrate intake. Int J Sports Med. 1998 Jun;19 Suppl 2:S142-5. doi: 10.1055/s-2007-971981. PMID 9694422
- [Result] Upshaw AU, Wong TS, Bandegan A, Lemon PW. Cycling Time Trial Performance 4 Hours After Glycogen-Lowering Exercise Is Similarly Enhanced by Recovery Nondairy Chocolate Beverages Versus Chocolate Milk. Int J Sport Nutr Exerc Metab. 2016 Feb;26(1):65-70. doi: 10.1123/ijsnem.2015-0056. Epub 2015 Aug 27. PMID 26314086